CLINICAL TRIAL: NCT01856192
Title: Randomized Phase II Open Label Study of Lenalidomide R-CHOP (R2CHOP) vs. RCHOP (Rituximab, Cyclophosphamide, Doxorubicin, Vincristine and Prednisone) in Patients With Newly Diagnosed Diffuse Large B Cell Lymphoma
Brief Title: Rituximab and Combination Chemotherapy With or Without Lenalidomide in Treating Patients With Newly Diagnosed Stage II-IV Diffuse Large B Cell Lymphoma
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2013-00959; NCI-2013-00959 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); ECOG-E1412; S13-01316; E1412; E1412 (Other: ECOG-ACRIN Cancer Research Group); E1412 (Other: CTEP); U10CA021115 (NIH); U10CA180820 (NIH); U24CA196172 (NIH)
Record Dates: First submitted 2013-05-14; First posted 2013-05-17 (Estimated); Results first posted 2021-06-03 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-10

CONDITIONS: Ann Arbor Stage II Diffuse Large B-Cell Lymphoma; Ann Arbor Stage III Diffuse Large B-Cell Lymphoma; Ann Arbor Stage IV Diffuse Large B-Cell Lymphoma
MeSH Terms: interventions — Cyclophosphamide; Doxorubicin; Lenalidomide; Prednisone; deltacortene; prednylidene; Rituximab; CT-P10; Vincristine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm A (rituximab, combination chemotherapy, lenalidomide) (Experimental): Patients receive rituximab IV, cyclophosphamide IV, doxorubicin hydrochloride IV, and vincristine sulfate IV on day 1; prednisone PO on days 1-5; and lenalidomide PO on days 1-10. Treatment repeats every 21 days for 6 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Cyclophosphamide; Drug: Doxorubicin Hydrochloride; Other: Laboratory Biomarker Analysis; Drug: Lenalidomide; Drug: Prednisone; Biological: Rituximab; Drug: Vincristine Sulfate
- Arm B (rituximab, combination chemotherapy) (Active Comparator): Patients receive rituximab, cyclophosphamide, doxorubicin hydrochloride, vincristine sulfate, and prednisone as in Arm A. Treatment repeats every 21 days for 6 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Cyclophosphamide; Drug: Doxorubicin Hydrochloride; Other: Laboratory Biomarker Analysis; Drug: Prednisone; Biological: Rituximab; Drug: Vincristine Sulfate

INTERVENTIONS:
Drug: Cyclophosphamide — Given IV
  Other Names: (-)-Cyclophosphamide; 2H-1,3,2-Oxazaphosphorine, 2-[bis(2-chloroethyl)amino]tetrahydro-, 2-oxide, monohydrate; Asta B 518; B 518; B-518; B518; Carloxan; Ciclofosfamida; Ciclofosfamide; Cicloxal; Clafen; Claphene; CP monohydrate; CTX; CYCLO-cell; Cycloblastin; Cycloblastine; Cyclophospham; Cyclophosphamid monohydrate; Cyclophosphamide Monohydrate; Cyclophosphamidum; Cyclophosphan; Cyclophosphane; Cyclophosphanum; Cyclostin; Cyclostine; Cytophosphan; Cytophosphane; Cytoxan; Fosfaseron; Genoxal; Genuxal; Ledoxina; Mitoxan; Neosar; Revimmune; Syklofosfamid; WR 138719; WR- 138719; WR-138719; WR138719
Drug: Doxorubicin Hydrochloride — Given IV
  Other Names: 5,12-Naphthacenedione, 10-[(3-amino-2,3,6-trideoxy-alpha-L-lyxo-hexopyranosyl)oxy]-7,8, 9,10-tetrahydro-6,8,11-trihydroxy-8-(hydroxyacetyl)-1-methoxy-, hydrochloride, (8S-cis)- (9CI); ADM; Adriacin; Adriamycin; Adriamycin Hydrochloride; Adriamycin PFS; Adriamycin RDF; ADRIAMYCIN, HYDROCHLORIDE; Adriamycine; Adriblastina; Adriblastine; Adrimedac; Chloridrato de Doxorrubicina; DOX; DOXO-CELL; Doxolem; Doxorubicin HCl; Doxorubicin.HCl; Doxorubin; Farmiblastina; FI 106; FI-106; FI106; hydroxydaunorubicin; Rubex
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Lenalidomide — Given PO
  Other Names: CC 5013; CC-5013; CC5013; CDC 501; Revlimid
  Arms: Arm A (rituximab, combination chemotherapy, lenalidomide)
Drug: Prednisone — Given PO
  Other Names: .delta.1-Cortisone; 1, 2-Dehydrocortisone; Adasone; Cortancyl; Dacortin; DeCortin; Decortisyl; Decorton; Delta 1-Cortisone; Delta-Dome; Deltacortene; Deltacortisone; Deltadehydrocortisone; Deltasone; Deltison; Deltra; Econosone; Lisacort; Meprosona-F; Metacortandracin; Meticorten; Ofisolona; Orasone; Panafcort; Panasol-S; Paracort; Perrigo Prednisone; PRED; Predicor; Predicorten; Prednicen-M; Prednicort; Prednidib; Prednilonga; Predniment; Prednisone Intensol; Prednisonum; Prednitone; Promifen; Rayos; Servisone; SK-Prednisone
Biological: Rituximab — Given IV
  Other Names: ABP 798; ABP-798; ABP798; BI 695500; BI-695500; BI695500; Blitzima; C2B8 Monoclonal Antibody; Chimeric Anti-CD20 Antibody; CT P10; CT-P10; CTP10; GP 2013; GP-2013; GP2013; IDEC 102; IDEC-102; IDEC-C2B8; IDEC-C2B8 Monoclonal Antibody; IDEC102; Ikgdar; Mabtas; MabThera; Monoclonal Antibody IDEC-C2B8; PF 05280586; PF-05280586; PF05280586; Riabni; Ritemvia; Rituxan; Rituximab ABBS; Rituximab ARRX; Rituximab Biosimilar ABP 798; Rituximab Biosimilar BI 695500; Rituximab Biosimilar CT-P10; Rituximab Biosimilar GB241; Rituximab Biosimilar GP2013; Rituximab Biosimilar IBI301; Rituximab Biosimilar JHL1101; Rituximab Biosimilar PF-05280586; Rituximab Biosimilar RTXM83; Rituximab Biosimilar SAIT101; Rituximab Biosimilar SIBP-02; rituximab biosimilar TQB2303; Rituximab PVVR; Rituximab-abbs; Rituximab-arrx; Rituximab-blit; Rituximab-pvvr; Rituximab-rite; Rituximab-rixa; Rituximab-rixi; Rixathon; Riximyo; RTXM 83; RTXM-83; RTXM83; Ruxience; Truxima
Drug: Vincristine Sulfate — Given IV
  Other Names: Kyocristine; Leurocristine Sulfate; Leurocristine, sulfate; Oncovin; Vincasar; Vincosid; Vincrex; Vincristine, sulfate

SUMMARY:
This randomized phase II trial studies how well rituximab and combination chemotherapy with or without lenalidomide work in treating patients with newly diagnosed stage II-IV diffuse large B cell lymphoma. Monoclonal antibodies, such as rituximab, may interfere with the ability of cancer cells to grow and spread. Drugs used in chemotherapy, such as cyclophosphamide, doxorubicin hydrochloride, vincristine sulfate, and prednisone, work in different ways to stop the growth of cancer cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Lenalidomide may stimulate the immune system in different ways and stop cancer cells from growing. It is not yet known whether rituximab and combination chemotherapy are more effective when given with or without lenalidomide in treating patients with diffuse large B cell lymphoma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Progression-free survival (PFS).

SECONDARY OBJECTIVES:

I. Response rate (RR). II. Complete remission (CR) rate as defined by positron emission tomography (PET)-computed tomography (CT) criteria.

III. Overall survival (OS).

TERTIARY OBJECTIVES:

I. Impact of diffuse large B cell lymphoma (DLBCL) molecular subtype on outcome.

II. Interim PET scan results in relation to treatment outcome.

OUTLINE: Patients are randomized to 1 of 2 treatment arms.

ARM A: Patients receive rituximab intravenously (IV), cyclophosphamide IV, doxorubicin hydrochloride IV, and vincristine sulfate IV on day 1; prednisone orally (PO) on days 1-5; and lenalidomide PO on days 1-10. Treatment repeats every 21 days for 6 courses in the absence of disease progression or unacceptable toxicity.

ARM B: Patients receive rituximab, cyclophosphamide, doxorubicin hydrochloride, vincristine sulfate, and prednisone as in Arm A. Treatment repeats every 21 days for 6 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3 months for 2 years, every 6 months for 1 year, and then annually for up to 7 years.

ELIGIBILITY:
Inclusion Criteria:

* PRE-REGISTRATION (STEP 0)
* Histologically confirmed DLBCL expressing CD20 antigen; patients with transformed lymphoma are excluded; in this regard, patients with composite lymphoma in the diagnostic tissue (concomitant DLBCL and follicular or other low-grade lymphoma component) are excluded; however, patients with DLBCL in primary diagnostic tissue but a bone marrow that shows low grade or indeterminate lymphoma are eligible; patients with known primary mediastinal large B-cell lymphoma (PMLBCL) are excluded; similarly, patients with known c-myc translocation (by fluorescence in situ hybridization) positive DLBCL are encouraged to participate in trials specifically designed for these patients; however patients with known c-myc DLBC positive are NOT excluded from this study; c-myc testing prior to study enrollment is NOT required
* Stages II bulky disease (defined as mass size of more than 10 cm), stage III, or IV (Ann Arbor staging); patients with stage I and stage II non-bulky disease are excluded from this study
* A paraffin-embedded tumor tissue specimen from the initial diagnostic biopsy has been located and ready to ship to the Mayo Clinic Lymphoma Laboratory following pre-registration; Note: excisional tumor biopsy is preferred; core needle biopsies will be considered adequate if there is enough tissue for the mandatory central pathology review immunohistochemistry and Genomics Education Partnership (GEP); submission of a tumor block is preferred, but if unavailable submit alternative materials
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2
* Previously untreated and not receiving any other agent that would be considered as a treatment for the lymphoma; for subjects with severe systemic symptoms, compressive disease, or rapidly progressing symptomatic adenopathy, are allowed for lymphoma associated symptom treatment with up to 1 mg/kg/day prednisone, or equivalent, for a maximum of 7 days is permitted prior to beginning the treatment, at the discretion of the investigator; a washout period does not apply
* No known central nervous system (CNS) lymphoma or cerebrospinal fluid involvement with malignant lymphoma cells; these patients are usually treated with CNS directed therapy; screening for cerebrospinal fluid (CSF)/CNS involvement is NOT required but can be performed per treating medical doctor (MD) discretion; intrathecal (IT) methotrexate or IT cytarabine prophylaxis in patients with negative CSF who are felt to be at high risk of CNS relapse is allowed per local MD discretion; this should be noted on the treatment form
* Absence of history of myocardial infarction =< 6 months, or congestive heart failure requiring use of ongoing maintenance therapy for life-threatening ventricular arrhythmias
* Absence of history of deep venous thrombosis/embolism, threatening thromboembolism or known thrombophilia; patients with a history of deep vein thrombosis(DVT)/pulmonary embolism (PE) or thrombophilia may participate if they are willing to be on full anticoagulation during the treatment if randomized to rituximab, cyclophosphamide, doxorubicin hydrochloride, vincristine sulfate, and prednisone (R2CHOP) arm A; full anticoagulation is defined as warfarin, factor X inhibitors, or low molecular weight heparin at therapeutic doses
* Patient must be able and willing to receive anticoagulation therapy with aspirin 70-325 mg daily prophylaxis, low molecular weight heparin, factor X inhibitors or warfarin; patients unable or unwilling to take any prophylaxis are NOT eligible
* Absence of history of acquired immune deficiency syndrome (AIDS)-related conditions (other than the presenting DLBCL) or post-transplant lymphoproliferative disorder (PTLD) in immunocompromised patients; patients with human immunodeficiency virus (HIV) on antiretroviral therapy other than zidovudine (AZT) and/or stavudine and without prior AIDS defining conditions and adequate CD4 count (> 400) are eligible
* No other active malignancy requiring therapy such as radiation, chemotherapy, or immunotherapy; exceptions to this are as follows: localized non-melanotic skin cancer and any cancer that in the judgment of the investigator has been treated with curative intent and will not interfere with the study treatment plan and response assessment
* No history of radiation therapy to >= 25% of the bone marrow for other diseases or history of anthracycline therapy
* Patients must not be receiving erythroid stimulating agents (EPO: Procrit, Aranesp)
* RANDOMIZATION (STEP 1)
* Patient meets the eligibility criteria outlined above
* Site has received notification from Mayo Clinic - Rochester Division of Hematopathology of the central confirmation of diagnosis and tissue adequacy for mandatory research studies
* Patients must have measurable disease (at least 1 lesion of >= 1.5 cm in one diameter) as detected by computed tomography (CT) or the CT images of the positron emission tomography (PET)/CT
* International Prognostic Index (IPI) of 2 or greater
* Ejection fraction of >= 45% by either multi-gated acquisition (MUGA) scan or echocardiogram (ECHO)
* Absence of co-morbid systemic illnesses or other severe concurrent disease which, in the judgment of the investigator, would make the patient inappropriate for entry into this study or interfere significantly with the proper assessment of safety and toxicity of the prescribed regimens, including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Absolute neutrophil count (ANC) >= 1500
* Platelets (PLT) >= 100,000
* Total bilirubin =< 1.5 x upper limit of normal (ULN) or if total bilirubin is > 1.5 x ULN, the direct bilirubin must be normal
* Alkaline (Alk.) phosphatase =< 3 x ULN unless evidence of the direct liver involvement by lymphoma - then =< 5 x ULN
* Aspartate aminotransferase (AST) =< 3 x ULN unless evidence of the direct liver involvement by lymphoma - then =< 5 x ULN
* Creatinine =< 2 x ULN or creatinine clearance (CrCl) > 30 ml/min
* Women must not be pregnant or breast-feeding
* Females of childbearing potential (FCBP) must have a negative serum or urine pregnancy test with a sensitivity of at least 25 mIU/mL within 10-14 days prior to and again within 24 hours of starting lenalidomide and must either commit to continued abstinence from heterosexual intercourse or begin TWO acceptable methods of birth control, one highly effective method and one additional effective method AT THE SAME TIME, at least 28 days before she starts taking lenalidomide; FCBP must also agree to ongoing pregnancy testing; a female of childbearing potential is any woman, regardless of sexual orientation or whether they have undergone tubal ligation, who meets the following criteria: 1) has not undergone a hysterectomy or bilateral oophorectomy; or 2) has not been naturally postmenopausal for at least 24 consecutive months (i.e., has had menses at any time in the preceding 24 consecutive months)
* Men must agree to use a latex condom during sexual contact with a FCBP even if they have had a successful vasectomy; all patients must be counseled at a minimum of every 28 days about pregnancy precautions and risks of fetal exposure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 349 (Actual)
Dates: Start 2013-08-27 (Actual); Primary Completion 2020-03-26 (Actual); Study Completion 2025-12-31 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Grzegorz S Nowakowski, Principal Investigator — ECOG-ACRIN Cancer Research Group
Locations (502):
- United States (502):
  - Alaska Breast Care and Surgery LLC, Anchorage, Alaska
  - Alaska Women's Cancer Care, Anchorage, Alaska
  - Anchorage Oncology Centre, Anchorage, Alaska
  - Katmai Oncology Group, Anchorage, Alaska
  - Providence Alaska Medical Center, Anchorage, Alaska
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - Banner University Medical Center - Tucson, Tucson, Arizona
  - University of Arizona Cancer Center-North Campus, Tucson, Arizona
  - John L McClellan Memorial Veterans Hospital, Little Rock, Arkansas
  - Kaiser Permanente-Deer Valley Medical Center, Antioch, California
  - Sutter Auburn Faith Hospital, Auburn, California
  - Kaiser Permanente-Baldwin Park, Baldwin Park, California
  - Kaiser Permanente-Bellflower, Bellflower, California
  - Providence Saint Joseph Medical Center/Disney Family Cancer Center, Burbank, California
  - Kaiser Permanente South Bay, Harbor City, California
  - Kaiser Permanente-Irvine, Irvine, California
  - Loma Linda University Medical Center, Loma Linda, California
  - Memorial Medical Center, Modesto, California
  - Palo Alto Medical Foundation-Camino Division, Mountain View, California
  - Palo Alto Medical Foundation-Gynecologic Oncology, Mountain View, California
  - Kaiser Permanente-Oakland, Oakland, California
  - UC Irvine Health/Chao Family Comprehensive Cancer Center, Orange, California
  - Palo Alto Medical Foundation Health Care, Palo Alto, California
  - Stanford Cancer Institute Palo Alto, Palo Alto, California
  - Kaiser Permanente - Panorama City, Panorama City, California
  - Kaiser Permanente-Richmond, Richmond, California
  - Sutter Medical Center Sacramento, Sacramento, California
  - Kaiser Permanente-South Sacramento, Sacramento, California
  - Kaiser Permanente Sacramento Medical Center, Sacramento, California
  - Kaiser Permanente-San Diego Mission, San Diego, California
  - Kaiser Permanente-San Diego Zion, San Diego, California
  - California Pacific Medical Center-Pacific Campus, San Francisco, California
  - Kaiser Permanente-San Francisco, San Francisco, California
  - Kaiser Permanente-Santa Teresa-San Jose, San Jose, California
  - Stanford Cancer Center South Bay, San Jose, California
  - Kaiser Permanente-San Marcos, San Marcos, California
  - Kaiser Permanente-San Rafael, San Rafael, California
  - Kaiser Permanente Medical Center - Santa Clara, Santa Clara, California
  - Palo Alto Medical Foundation-Santa Cruz, Santa Cruz, California
  - Kaiser Permanente-Santa Rosa, Santa Rosa, California
  - Sutter Pacific Medical Foundation, Santa Rosa, California
  - Kaiser Permanente-South San Francisco, South San Francisco, California
  - Palo Alto Medical Foundation-Sunnyvale, Sunnyvale, California
  - Kaiser Permanente-Walnut Creek, Walnut Creek, California
  - Kaiser Permanente-Woodland Hills, Woodland Hills, California
  - Rocky Mountain Cancer Centers-Aurora, Aurora, Colorado
  - The Medical Center of Aurora, Aurora, Colorado
  - Boulder Community Foothills Hospital, Boulder, Colorado
  - Penrose-Saint Francis Healthcare, Colorado Springs, Colorado
  - Rocky Mountain Cancer Centers-Penrose, Colorado Springs, Colorado
  - Kaiser Permanente-Franklin, Denver, Colorado
  - AdventHealth Porter, Denver, Colorado
  - Colorado Blood Cancer Institute, Denver, Colorado
  - Presbyterian - Saint Lukes Medical Center - Health One, Denver, Colorado
  - Rocky Mountain Cancer Centers-Midtown, Denver, Colorado
  - Saint Joseph Hospital - Cancer Centers of Colorado, Denver, Colorado
  - Rocky Mountain Cancer Centers-Rose, Denver, Colorado
  - Rose Medical Center, Denver, Colorado
  - Western States Cancer Research NCORP, Denver, Colorado
  - Mercy Medical Center, Durango, Colorado
  - Mountain Blue Cancer Care Center - Swedish, Englewood, Colorado
  - Swedish Medical Center, Englewood, Colorado
  - Mountain Blue Cancer Care Center, Golden, Colorado
  - Banner North Colorado Medical Center, Greeley, Colorado
  - Rocky Mountain Cancer Centers-Greenwood Village, Greenwood Village, Colorado
  - Kaiser Permanente-Rock Creek, Lafayette, Colorado
  - Rocky Mountain Cancer Centers-Lakewood, Lakewood, Colorado
  - Saint Anthony Hospital, Lakewood, Colorado
  - Rocky Mountain Cancer Centers-Littleton, Littleton, Colorado
  - AdventHealth Littleton, Littleton, Colorado
  - Rocky Mountain Cancer Centers-Sky Ridge, Lone Tree, Colorado
  - Sky Ridge Medical Center, Lone Tree, Colorado
  - Longmont United Hospital, Longmont, Colorado
  - Rocky Mountain Cancer Centers-Longmont, Longmont, Colorado
  - Banner North Colorado Medical Center - Loveland Campus, Loveland, Colorado
  - AdventHealth Parker, Parker, Colorado
  - Rocky Mountain Cancer Centers-Parker, Parker, Colorado
  - Saint Mary Corwin Medical Center, Pueblo, Colorado
  - Rocky Mountain Cancer Centers-Thornton, Thornton, Colorado
  - Intermountain Health Lutheran Hospital, Wheat Ridge, Colorado
  - Smilow Cancer Hospital Care Center at Saint Francis, Hartford, Connecticut
  - The Hospital of Central Connecticut, New Britain, Connecticut
  - Yale University, New Haven, Connecticut
  - Bayhealth Hospital Kent Campus, Dover, Delaware
  - Beebe Medical Center, Lewes, Delaware
  - Delaware Clinical and Laboratory Physicians PA, Newark, Delaware
  - Helen F Graham Cancer Center, Newark, Delaware
  - Medical Oncology Hematology Consultants PA, Newark, Delaware
  - Christiana Care Health System-Christiana Hospital, Newark, Delaware
  - Beebe Health Campus, Rehoboth Beach, Delaware
  - TidalHealth Nanticoke / Allen Cancer Center, Seaford, Delaware
  - Sibley Memorial Hospital, Washington D.C., District of Columbia
  - The Watson Clinic, Lakeland, Florida
  - Orlando Health Cancer Institute, Orlando, Florida
  - Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia
  - Northside Hospital, Atlanta, Georgia
  - Atlanta VA Medical Center, Decatur, Georgia
  - Northside Hospital - Gwinnett, Lawrenceville, Georgia
  - Atrium Health Navicent, Macon, Georgia
  - Lewis Cancer and Research Pavilion at Saint Joseph's/Candler, Savannah, Georgia
  - Hawaii Cancer Care Inc - Waterfront Plaza, Honolulu, Hawaii
  - Straub Clinic and Hospital, Honolulu, Hawaii
  - University of Hawaii Cancer Center, Honolulu, Hawaii
  - Queen's Cancer Center - Kuakini, Honolulu, Hawaii
  - The Cancer Center of Hawaii-Liliha, Honolulu, Hawaii
  - Kaiser Permanente Moanalua Medical Center, Honolulu, Hawaii
  - Saint Alphonsus Cancer Care Center-Boise, Boise, Idaho
  - Saint Luke's Cancer Institute - Boise, Boise, Idaho
  - Saint Luke's Cancer Institute - Fruitland, Fruitland, Idaho
  - Saint Luke's Cancer Institute - Meridian, Meridian, Idaho
  - Saint Luke's Cancer Institute - Nampa, Nampa, Idaho
  - Kootenai Clinic Cancer Services - Post Falls, Post Falls, Idaho
  - Saint Luke's Cancer Institute - Twin Falls, Twin Falls, Idaho
  - Illinois CancerCare-Bloomington, Bloomington, Illinois
  - Illinois CancerCare-Canton, Canton, Illinois
  - Illinois CancerCare-Carthage, Carthage, Illinois
  - Northwestern University, Chicago, Illinois
  - Weiss Memorial Hospital, Chicago, Illinois
  - UChicago Medicine Comprehensive Cancer Center - Saint Joseph Hospital, Chicago, Illinois
  - Carle at The Riverfront, Danville, Illinois
  - Cancer Care Specialists of Illinois - Decatur, Decatur, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Heartland Cancer Research NCORP, Decatur, Illinois
  - Carle Physician Group-Effingham, Effingham, Illinois
  - Crossroads Cancer Center, Effingham, Illinois
  - Ascension Alexian Brothers - Elk Grove Village, Elk Grove Village, Illinois
  - Illinois CancerCare-Eureka, Eureka, Illinois
  - Illinois CancerCare-Galesburg, Galesburg, Illinois
  - Northwestern Medicine Cancer Center Delnor, Geneva, Illinois
  - Ingalls Memorial Hospital, Harvey, Illinois
  - Hinsdale Hematology Oncology Associates Incorporated, Hinsdale, Illinois
  - Duly Health and Care Joliet, Joliet, Illinois
  - Illinois CancerCare-Kewanee Clinic, Kewanee, Illinois
  - Illinois CancerCare-Macomb, Macomb, Illinois
  - Carle Physician Group-Mattoon/Charleston, Mattoon, Illinois
  - Trinity Medical Center, Moline, Illinois
  - Illinois CancerCare-Monmouth, Monmouth, Illinois
  - Illinois Cancer Specialists-Niles, Niles, Illinois
  - Cancer Care Center of O'Fallon, O'Fallon, Illinois
  - Illinois CancerCare-Ottawa Clinic, Ottawa, Illinois
  - Illinois CancerCare-Pekin, Pekin, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - Illinois CancerCare-Peru, Peru, Illinois
  - Illinois CancerCare-Princeton, Princeton, Illinois
  - West Suburban Medical Center, River Forest, Illinois
  - Swedish American Hospital, Rockford, Illinois
  - UW Health Carbone Cancer Center Rockford, Rockford, Illinois
  - Central Illinois Hematology Oncology Center, Springfield, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Springfield Clinic, Springfield, Illinois
  - Springfield Memorial Hospital, Springfield, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - The Carle Foundation Hospital, Urbana, Illinois
  - Northwestern Medicine Cancer Center Warrenville, Warrenville, Illinois
  - Elkhart Clinic, Elkhart, Indiana
  - Michiana Hematology Oncology PC-Elkhart, Elkhart, Indiana
  - Elkhart General Hospital, Elkhart, Indiana
  - Indiana University/Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - IU Health Central Indiana Cancer Centers-East, Indianapolis, Indiana
  - Community Howard Regional Health, Kokomo, Indiana
  - IU Health La Porte Hospital, La Porte, Indiana
  - IU Health Arnett Cancer Care, Lafayette, Indiana
  - Premier Oncology Hematology Associates, Merrillville, Indiana
  - Michiana Hematology Oncology PC-Mishawaka, Mishawaka, Indiana
  - Saint Joseph Regional Medical Center-Mishawaka, Mishawaka, Indiana
  - IU Health Ball Memorial Hospital, Muncie, Indiana
  - Michiana Hematology Oncology PC-Plymouth, Plymouth, Indiana
  - Reid Health, Richmond, Indiana
  - Northern Indiana Cancer Research Consortium, South Bend, Indiana
  - Michiana Hematology Oncology PC-Westville, Westville, Indiana
  - McFarland Clinic - Ames, Ames, Iowa
  - Oncology Associates at Mercy Medical Center, Cedar Rapids, Iowa
  - Mercy Cancer Center-West Lakes, Clive, Iowa
  - UI Health Care Mission Cancer and Blood - West Des Moines Clinic, Clive, Iowa
  - Iowa-Wide Oncology Research Coalition NCORP, Des Moines, Iowa
  - UI Health Care Mission Cancer and Blood - Des Moines Clinic, Des Moines, Iowa
  - Mercy Medical Center - Des Moines, Des Moines, Iowa
  - UI Health Care Mission Cancer and Blood - Laurel Clinic, Des Moines, Iowa
  - Mercy Medical Center - North Iowa, Mason City, Iowa
  - Ottumwa Regional Health Center, Ottumwa, Iowa
  - Siouxland Regional Cancer Center, Sioux City, Iowa
  - MercyOne Waterloo Cancer Center, Waterloo, Iowa
  - Mercy Medical Center-West Lakes, West Des Moines, Iowa
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - Kansas City NCI Community Oncology Research Program, Prairie Village, Kansas
  - Wesley Medical Center, Wichita, Kansas
  - Flaget Memorial Hospital, Bardstown, Kentucky
  - Jewish Hospital, Louisville, Kentucky
  - UofL Health Medical Center Northeast, Louisville, Kentucky
  - Ochsner Health Center-Summa, Baton Rouge, Louisiana
  - Ochsner Medical Center Kenner, Kenner, Louisiana
  - Ochsner LSU Health Monroe Medical Center, Monroe, Louisiana
  - Ochsner Medical Center Jefferson, New Orleans, Louisiana
  - LSU Health Sciences Center at Shreveport, Shreveport, Louisiana
  - Harold Alfond Center for Cancer Care, Augusta, Maine
  - Eastern Maine Medical Center, Bangor, Maine
  - Lafayette Family Cancer Center-EMMC, Brewer, Maine
  - Greater Baltimore Medical Center, Baltimore, Maryland
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - Christiana Care - Union Hospital, Elkton, Maryland
  - TidalHealth Peninsula Regional, Salisbury, Maryland
  - Tufts Medical Center, Boston, Massachusetts
  - Boston Medical Center, Boston, Massachusetts
  - Baystate Medical Center, Springfield, Massachusetts
  - UMass Memorial Medical Center - University Campus, Worcester, Massachusetts
  - Trinity Health Saint Joseph Mercy Hospital Ann Arbor, Ann Arbor, Michigan
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Bronson Battle Creek, Battle Creek, Michigan
  - Corewell Health Dearborn Hospital, Dearborn, Michigan
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Henry Ford Health Saint John Hospital, Detroit, Michigan
  - OSF Saint Francis Hospital and Medical Group, Escanaba, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Corewell Health Grand Rapids Hospitals - Butterworth Hospital, Grand Rapids, Michigan
  - Trinity Health Grand Rapids Hospital, Grand Rapids, Michigan
  - Allegiance Health, Jackson, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Trinity Health Saint Mary Mercy Livonia Hospital, Livonia, Michigan
  - Trinity Health Muskegon Hospital, Muskegon, Michigan
  - Trinity Health Saint Joseph Mercy Oakland Hospital, Pontiac, Michigan
  - Lake Huron Medical Center, Port Huron, Michigan
  - Corewell Health Reed City Hospital, Reed City, Michigan
  - MyMichigan Medical Center Saginaw, Saginaw, Michigan
  - Corewell Health Lakeland Hospitals - Marie Yeager Cancer Center, Saint Joseph, Michigan
  - Corewell Health Lakeland Hospitals - Saint Joseph Hospital, Saint Joseph, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - Henry Ford Health Warren Hospital, Warren, Michigan
  - Sanford Joe Lueken Cancer Center, Bemidji, Minnesota
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Mercy Hospital, Coon Rapids, Minnesota
  - Essentia Health Cancer Center, Duluth, Minnesota
  - Saint Luke's Hospital of Duluth, Duluth, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Lake Region Healthcare Corporation-Cancer Care, Fergus Falls, Minnesota
  - Unity Hospital, Fridley, Minnesota
  - Hutchinson Area Health Care, Hutchinson, Minnesota
  - Minnesota Oncology Hematology PA-Maplewood, Maplewood, Minnesota
  - Saint John's Hospital - Healtheast, Maplewood, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - Health Partners Inc, Minneapolis, Minnesota
  - North Memorial Medical Health Center, Robbinsdale, Minnesota
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - Coborn Cancer Center at Saint Cloud Hospital, Saint Cloud, Minnesota
  - Metro Minnesota Community Oncology Research Consortium, Saint Louis Park, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Saint Francis Regional Medical Center, Shakopee, Minnesota
  - Lakeview Hospital, Stillwater, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Rice Memorial Hospital, Willmar, Minnesota
  - Minnesota Oncology Hematology PA-Woodbury, Woodbury, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Central Care Cancer Center - Bolivar, Bolivar, Missouri
  - Mercy Cancer Center - Cape Girardeau, Cape Girardeau, Missouri
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - Saint Luke's Hospital, Chesterfield, Missouri
  - MU Health Care Goldschmidt Cancer Center, Jefferson City, Missouri
  - Saint Luke's Hospital of Kansas City, Kansas City, Missouri
  - Mercy Clinic-Rolla-Cancer and Hematology, Rolla, Missouri
  - Phelps Health Delbert Day Cancer Institute, Rolla, Missouri
  - Mercy Hospital Springfield, Springfield, Missouri
  - CoxHealth South Hospital, Springfield, Missouri
  - Mercy Infusion Center - Chippewa, St Louis, Missouri
  - Missouri Baptist Medical Center, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Billings Clinic Cancer Center, Billings, Montana
  - Bozeman Health Deaconess Hospital, Bozeman, Montana
  - Saint James Community Hospital and Cancer Treatment Center, Butte, Montana
  - Benefis Sletten Cancer Institute, Great Falls, Montana
  - Logan Health Medical Center, Kalispell, Montana
  - Saint Patrick Hospital - Community Hospital, Missoula, Montana
  - Community Medical Center, Missoula, Montana
  - Nebraska Cancer Specialists/Oncology Hematology West PC, Grand Island, Nebraska
  - CHI Health Good Samaritan, Kearney, Nebraska
  - Nebraska Hematology and Oncology, Lincoln, Nebraska
  - Nebraska Cancer Research Center, Lincoln, Nebraska
  - Cancer Partners of Nebraska, Lincoln, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Cancer and Blood Specialists-Henderson, Henderson, Nevada
  - Comprehensive Cancer Centers of Nevada - Henderson, Henderson, Nevada
  - Las Vegas Cancer Center-Henderson, Henderson, Nevada
  - Comprehensive Cancer Centers of Nevada-Southeast Henderson, Henderson, Nevada
  - Oncology Las Vegas - Henderson, Henderson, Nevada
  - University Medical Center of Southern Nevada, Las Vegas, Nevada
  - Cancer and Blood Specialists-Shadow, Las Vegas, Nevada
  - Radiation Oncology Centers of Nevada Central, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-Maryland Parkway, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-San Martin, Las Vegas, Nevada
  - Radiation Oncology Centers of Nevada Southeast, Las Vegas, Nevada
  - Nevada Cancer Research Foundation NCORP, Las Vegas, Nevada
  - Cancer Therapy and Integrative Medicine, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada - Northwest, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-Tenaya, Las Vegas, Nevada
  - Oncology Las Vegas - Tenaya, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada-Summerlin, Las Vegas, Nevada
  - Las Vegas Cancer Center-Medical Center, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - OptumCare Cancer Care at Fort Apache, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-Centennial Hills, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada - Central Valley, Las Vegas, Nevada
  - New Hampshire Oncology Hematology PA-Concord, Concord, New Hampshire
  - Wentworth-Douglass Hospital, Dover, New Hampshire
  - LRGHealthcare-Lakes Region General Hospital, Laconia, New Hampshire
  - Dartmouth Hitchcock Medical Center/Dartmouth Cancer Center, Lebanon, New Hampshire
  - Solinsky Center for Cancer Care, Manchester, New Hampshire
  - Cooper Hospital University Medical Center, Camden, New Jersey
  - Englewood Hospital and Medical Center, Englewood, New Jersey
  - Saint Barnabas Medical Center, Livingston, New Jersey
  - Virtua Memorial, Mount Holly, New Jersey
  - Inspira Medical Center Mullica Hill, Mullica Hill, New Jersey
  - The Valley Hospital - Luckow Pavilion, Paramus, New Jersey
  - Valley Health System Ridgewood Campus, Ridgewood, New Jersey
  - Inspira Medical Center Vineland, Vineland, New Jersey
  - Valley Health System-Hematology/Oncology, Westwood, New Jersey
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Presbyterian Kaseman Hospital, Albuquerque, New Mexico
  - Memorial Medical Center-Las Cruces, Las Cruces, New Mexico
  - Christus Saint Vincent Regional Cancer Center, Santa Fe, New Mexico
  - Kings County Hospital, Brooklyn, New York
  - State University of New York Downstate Medical Center, Brooklyn, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - Hematology Oncology Associates of Central New York-East Syracuse, East Syracuse, New York
  - Laura and Isaac Perlmutter Cancer Center at NYU Langone, New York, New York
  - NYP/Columbia University Medical Center/Herbert Irving Comprehensive Cancer Center, New York, New York
  - Champlain Valley Physicians Hospital Medical Center, Plattsburgh, New York
  - University of Rochester, Rochester, New York
  - State University of New York Upstate Medical University, Syracuse, New York
  - Montefiore Medical Center-Einstein Campus, The Bronx, New York
  - Montefiore Medical Center-Weiler Hospital, The Bronx, New York
  - Montefiore Medical Center - Moses Campus, The Bronx, New York
  - Randolph Hospital, Asheboro, North Carolina
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Southeastern Medical Oncology Center-Clinton, Clinton, North Carolina
  - Southeastern Medical Oncology Center-Goldsboro, Goldsboro, North Carolina
  - Wayne Memorial Hospital, Goldsboro, North Carolina
  - Cone Health Cancer Center, Greensboro, North Carolina
  - Margaret R Pardee Memorial Hospital, Hendersonville, North Carolina
  - Southeastern Medical Oncology Center-Jacksonville, Jacksonville, North Carolina
  - ECU Health Oncology Kinston, Kinston, North Carolina
  - Annie Penn Memorial Hospital, Reidsville, North Carolina
  - Iredell Memorial Hospital, Statesville, North Carolina
  - Marion L Shepard Cancer Center - ECU Health Beaufort Hospital, Washington, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Sanford Bismarck Medical Center, Bismarck, North Dakota
  - Sanford Broadway Medical Center, Fargo, North Dakota
  - Sanford Roger Maris Cancer Center, Fargo, North Dakota
  - Summa Health System - Akron Campus, Akron, Ohio
  - Cleveland Clinic Akron General, Akron, Ohio
  - Summa Health System - Barberton Campus, Barberton, Ohio
  - Cleveland Clinic Mercy Hospital, Canton, Ohio
  - Geauga Hospital, Chardon, Ohio
  - University of Cincinnati Cancer Center-UC Medical Center, Cincinnati, Ohio
  - Good Samaritan Hospital - Cincinnati, Cincinnati, Ohio
  - TriHealth Cancer Institute-Westside, Cincinnati, Ohio
  - TriHealth Cancer Institute-Anderson, Cincinnati, Ohio
  - Case Western Reserve University, Cleveland, Ohio
  - MetroHealth Medical Center, Cleveland, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Columbus Oncology and Hematology Associates Inc, Columbus, Ohio
  - Riverside Methodist Hospital, Columbus, Ohio
  - Columbus NCI Community Oncology Research Program, Columbus, Ohio
  - The Mark H Zangmeister Center, Columbus, Ohio
  - Mount Carmel Health Center West, Columbus, Ohio
  - Good Samaritan Hospital - Dayton, Dayton, Ohio
  - Miami Valley Hospital, Dayton, Ohio
  - Miami Valley Hospital North, Dayton, Ohio
  - Mercy Cancer Center-Elyria, Elyria, Ohio
  - Blanchard Valley Hospital, Findlay, Ohio
  - Saint Rita's Medical Center, Lima, Ohio
  - Marietta Memorial Hospital, Marietta, Ohio
  - Toledo Clinic Cancer Centers-Maumee, Maumee, Ohio
  - UH Seidman Cancer Center at Landerbrook Health Center, Mayfield Heights, Ohio
  - UH Seidman Cancer Center at Lake Health Mentor Campus, Mentor, Ohio
  - Licking Memorial Hospital, Newark, Ohio
  - UH Seidman Cancer Center at Firelands Regional Medical Center, Sandusky, Ohio
  - Springfield Regional Cancer Center, Springfield, Ohio
  - Springfield Regional Medical Center, Springfield, Ohio
  - ProMedica Flower Hospital, Sylvania, Ohio
  - University of Toledo, Toledo, Ohio
  - Toledo Clinic Cancer Centers-Toledo, Toledo, Ohio
  - Saint Ann's Hospital, Westerville, Ohio
  - UH Seidman Cancer Center at Saint John Medical Center, Westlake, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Oklahoma Cancer Specialists and Research Institute-Tulsa, Tulsa, Oklahoma
  - Clackamas Radiation Oncology Center, Clackamas, Oregon
  - Providence Cancer Institute Clackamas Clinic, Clackamas, Oregon
  - Bay Area Hospital, Coos Bay, Oregon
  - Providence Newberg Medical Center, Newberg, Oregon
  - Providence Willamette Falls Medical Center, Oregon City, Oregon
  - Providence Portland Medical Center, Portland, Oregon
  - Providence Saint Vincent Medical Center, Portland, Oregon
  - Lehigh Valley Hospital-Cedar Crest, Allentown, Pennsylvania
  - Saint Luke's University Hospital-Bethlehem Campus, Bethlehem, Pennsylvania
  - Bryn Mawr Hospital, Bryn Mawr, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - Doylestown Hospital, Doylestown, Pennsylvania
  - Delaware County Memorial Hospital, Drexel Hill, Pennsylvania
  - Ephrata Cancer Center, Ephrata, Pennsylvania
  - Ephrata Community Hospital, Ephrata, Pennsylvania
  - Adams Cancer Center, Gettysburg, Pennsylvania
  - WellSpan Medical Oncology and Hematology, Hanover, Pennsylvania
  - Geisinger Medical Center-Cancer Center Hazleton, Hazleton, Pennsylvania
  - Penn State Milton S Hershey Medical Center, Hershey, Pennsylvania
  - Geisinger Medical Oncology-Lewisburg, Lewisburg, Pennsylvania
  - Paoli Memorial Hospital, Paoli, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Temple University Hospital, Philadelphia, Pennsylvania
  - Pottstown Hospital, Pottstown, Pennsylvania
  - Geisinger Cancer Services-Pottsville, Pottsville, Pennsylvania
  - Hematology and Oncology Associates of North East Pennsylvania, Scranton, Pennsylvania
  - Geisinger Medical Oncology-Selinsgrove, Selinsgrove, Pennsylvania
  - Grand View Hospital, Sellersville, Pennsylvania
  - Mount Nittany Medical Center, State College, Pennsylvania
  - Chester County Hospital, West Chester, Pennsylvania
  - Reading Hospital, West Reading, Pennsylvania
  - Geisinger Wyoming Valley/Henry Cancer Center, Wilkes-Barre, Pennsylvania
  - Lankenau Medical Center, Wynnewood, Pennsylvania
  - WellSpan Health-York Hospital, York, Pennsylvania
  - Prisma Health Cancer Institute - Spartanburg, Boiling Springs, South Carolina
  - Prisma Health Cancer Institute - Easley, Easley, South Carolina
  - Greenville Health System Cancer Institute-Andrews, Greenville, South Carolina
  - Prisma Health Cancer Institute - Butternut, Greenville, South Carolina
  - Prisma Health Cancer Institute - Faris, Greenville, South Carolina
  - Prisma Health Greenville Memorial Hospital, Greenville, South Carolina
  - Prisma Health Cancer Institute - Eastside, Greenville, South Carolina
  - Prisma Health Cancer Institute - Greer, Greer, South Carolina
  - Prisma Health Cancer Institute - Seneca, Seneca, South Carolina
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - Sanford Cancer Center Oncology Clinic, Sioux Falls, South Dakota
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - Dell Seton Medical Center at The University of Texas, Austin, Texas
  - Parkland Memorial Hospital, Dallas, Texas
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - Brooke Army Medical Center, Fort Sam Houston, Texas
  - Covenant Medical Center-Lakeside, Lubbock, Texas
  - Texas Tech University Health Sciences Center-Lubbock, Lubbock, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah
  - University of Virginia Cancer Center, Charlottesville, Virginia
  - Augusta Health Center for Cancer and Blood Disorders, Fishersville, Virginia
  - Sovah Health Martinsville, Martinsville, Virginia
  - Swedish Cancer Institute-Edmonds, Edmonds, Washington
  - PeaceHealth Saint John Medical Center, Longview, Washington
  - Swedish Medical Center-Ballard Campus, Seattle, Washington
  - Swedish Medical Center-First Hill, Seattle, Washington
  - PeaceHealth Southwest Medical Center, Vancouver, Washington
  - West Virginia University Charleston Division, Charleston, West Virginia
  - Langlade Hospital and Cancer Center, Antigo, Wisconsin
  - ThedaCare Regional Cancer Center, Appleton, Wisconsin
  - Aurora Cancer Care-Southern Lakes VLCC, Burlington, Wisconsin
  - HSHS Sacred Heart Hospital, Eau Claire, Wisconsin
  - Marshfield Clinic Cancer Center at Sacred Heart, Eau Claire, Wisconsin
  - Aurora Health Care Germantown Health Center, Germantown, Wisconsin
  - Aurora Cancer Care-Grafton, Grafton, Wisconsin
  - Green Bay Oncology at Saint Vincent Hospital, Green Bay, Wisconsin
  - Bellin Memorial Hospital, Green Bay, Wisconsin
  - Saint Vincent Hospital Cancer Center Green Bay, Green Bay, Wisconsin
  - Saint Vincent Hospital Cancer Center at Saint Mary's, Green Bay, Wisconsin
  - Aurora BayCare Medical Center, Green Bay, Wisconsin
  - University of Wisconsin Carbone Cancer Center - Johnson Creek, Johnson Creek, Wisconsin
  - Aurora Cancer Care-Kenosha South, Kenosha, Wisconsin
  - Gundersen Lutheran Medical Center, La Crosse, Wisconsin
  - SSM Health Dean Medical Group - South Madison Campus, Madison, Wisconsin
  - University of Wisconsin Carbone Cancer Center - University Hospital, Madison, Wisconsin
  - Holy Family Memorial Hospital, Manitowoc, Wisconsin
  - Aurora Bay Area Medical Group-Marinette, Marinette, Wisconsin
  - Bay Area Medical Center, Marinette, Wisconsin
  - Marshfield Medical Center-Marshfield, Marshfield, Wisconsin
  - Marshfield Medical Center, Marshfield, Wisconsin
  - Aurora Cancer Care-Milwaukee, Milwaukee, Wisconsin
  - Aurora Saint Luke's Medical Center, Milwaukee, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
  - Aurora Sinai Medical Center, Milwaukee, Wisconsin
  - Marshfield Medical Center - Minocqua, Minocqua, Wisconsin
  - Cancer Center of Western Wisconsin, New Richmond, Wisconsin
  - ProHealth Oconomowoc Memorial Hospital, Oconomowoc, Wisconsin
  - Saint Vincent Hospital Cancer Center at Oconto Falls, Oconto Falls, Wisconsin
  - Vince Lombardi Cancer Clinic - Oshkosh, Oshkosh, Wisconsin
  - Aurora Cancer Care-Racine, Racine, Wisconsin
  - Aspirus Cancer Care - James Beck Cancer Center, Rhinelander, Wisconsin
  - Saint Mary's Hospital, Rhinelander, Wisconsin
  - Lakeview Medical Center-Marshfield Clinic, Rice Lake, Wisconsin
  - Marshfield Medical Center-Rice Lake, Rice Lake, Wisconsin
  - Vince Lombardi Cancer Clinic-Sheboygan, Sheboygan, Wisconsin
  - Aspirus Cancer Care - Stevens Point, Stevens Point, Wisconsin
  - Aurora Medical Center in Summit, Summit, Wisconsin
  - Vince Lombardi Cancer Clinic-Two Rivers, Two Rivers, Wisconsin
  - Aurora Cancer Care-Waukesha, Waukesha, Wisconsin
  - ProHealth Waukesha Memorial Hospital, Waukesha, Wisconsin
  - UW Cancer Center at ProHealth Care, Waukesha, Wisconsin
  - Aspirus Regional Cancer Center, Wausau, Wisconsin
  - Marshfield Clinic-Wausau Center, Wausau, Wisconsin
  - Aurora Cancer Care-Milwaukee West, Wauwatosa, Wisconsin
  - Aurora West Allis Medical Center, West Allis, Wisconsin
  - Marshfield Medical Center - Weston, Weston, Wisconsin
  - Aspirus Cancer Care - Wisconsin Rapids, Wisconsin Rapids, Wisconsin
  - Marshfield Clinic - Wisconsin Rapids Center, Wisconsin Rapids, Wisconsin

REFERENCES:
- [Derived] King RL, Nowakowski GS, Witzig TE, Scott DW, Little RF, Hong F, Gascoyne RD, Kahl BS, Macon WR. Rapid, real time pathology review for ECOG/ACRIN 1412: a novel and successful paradigm for future lymphoma clinical trials in the precision medicine era. Blood Cancer J. 2018 Feb 28;8(3):27. doi: 10.1038/s41408-018-0064-9. PMID 29531316

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between August 2013 and January 2017, 349 patients were enrolled on this study.
Groups:
- Arm A (R2CHOP): Patients receive rituximab IV, cyclophosphamide IV, doxorubicin hydrochloride IV, and vincristine sulfate IV on day 1; prednisone PO on days 1-5; and lenalidomide PO on days 1-10. Treatment repeats every 21 days for 6 courses in the absence of disease progression or unacceptable toxicity.
- Arm B (RCHOP): Patients receive rituximab, cyclophosphamide, doxorubicin hydrochloride, vincristine sulfate, and prednisone as in Arm A. Treatment repeats every 21 days for 6 courses in the absence of disease progression or unacceptable toxicity.
Period: Overall Study
Arm/Group | Arm A (R2CHOP) | Arm B (RCHOP)
Started | 173 | 176
Treated Patients | 166 | 171
Evaluable Patients (Eligible and Treated) | 145 | 135
Completed | 124 | 116
Not Completed | 49 | 60
Not completed — Adverse Event | 12 | 4
Not completed — Alternative therapy | 0 | 3
Not completed — Death | 3 | 5
Not completed — Lack of Efficacy | 0 | 5
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Other diseases | 1 | 0
Not completed — Never started treatment | 7 | 5
Not completed — Path ineligible | 20 | 34
Not completed — Non-path ineligible | 2 | 2
Not completed — Physician Decision | 1 | 1
Not completed — Suspicion of progressive disease | 1 | 0
Not completed — Non-compliance | 1 | 0

BASELINE CHARACTERISTICS:
Population: All evaluable (treated and eligible) patients
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A (R2CHOP) | Arm B (RCHOP) | Total
Number analyzed (Participants) | 145 | 135 | 280
Age, Continuous [Median (Full Range); unit: years] | 67 [24 to 88] | 66 [37 to 92] | 66 [24 to 92]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 51 | 59 | 110
  Male | 94 | 76 | 170
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 5 | 8
  Not Hispanic or Latino | 137 | 125 | 262
  Unknown or Not Reported | 5 | 5 | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 6 | 2 | 8
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 10 | 16
  White | 128 | 118 | 246
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 5 | 5 | 10

OUTCOME MEASURES:

1. Primary Outcome: 3-year Progression-free Survival Rate
Description: Progression-free survival is defined as the time from randomization to disease progression, new primary of the same type or death, whichever occurs first. Progressive disease is defined as:
  * Appearance of any new lesion more than 1.5 cm in any axis during or at the end of therapy, even if other lesions are decreasing in size.
  * >= 50% increase from nadir in the sum of the product of the diameters of any previously involved nodes or extranodal masses, or in a single involved node or extranodal mass, or the size of other lesions.
  * >= 50% increase in the longest diameter of any single previously identified node or extranodal mass > 1 cm in its short axis.
  * Lesions should be PET positive unless the lesion is too small to be detected with current PET systems.
  * Measurable extranodal disease should be assessed in a manner similar to that for nodal disease.
    3-year progression-free survival rate was calculated using Kaplan-Meier method.
Time Frame: Assessed every 3 months for 2 years, every 6 months for year 3, and then annually for years 4-10, 3-year PFS rate reported
Population: Evaluable (eligible and treated) patients
Measure: Number (80% Confidence Interval); unit: proportion of participants
Arm/Group | Arm A (R2CHOP) | Arm B (RCHOP)
Number analyzed (Participants) | 145 | 135
proportion of participants | 0.727 [0.678 to 0.779] | 0.615 [0.562 to 0.674]
Statistical Analysis 1: Comparison: Arm A (R2CHOP) vs Arm B (RCHOP); Test type: Superiority; p = 0.03, Log Rank; Stratified log rank test

2. Secondary Outcome: Proportion of Patients With Response
Description: Response is defined as complete response (CR) or partial response (PR) CR: Complete disappearance of all detectable clinical evidence of disease and disease-related symptoms
  PR:
  * >=50% decrease in sum of the product of the diameters (SPD) of up to 6 of the largest dominant nodes or extranodal masses
  * No increase in the size of other nodes, liver or spleen
  * Bone marrow assessment is irrelevant for determination of a PR if the sample was positive prior to treatment. However, if positive, the cell type should be specified
  * No new sites of disease
  * The post-treatment PET should be positive at any previously involved sites
  * For variably FDG-avid lymphomas/FDG-avidity unknown, without a pretreatment PET scan, or if a pretreatment PET scan was negative, CT scan criteria should be used
  * Patients with a CR and persistent morphologic bone marrow involvement
  * Patients with bone marrow involved before therapy and a clinical CR but no bone marrow assessment after treatment
Time Frame: Assessed every 3 months for 2 years, every 6 months for year 3, and then annually for years 4-10
Population: Evaluable (eligible and treated) patients
Measure: Number (90% Confidence Interval); unit: proportion of participants
Arm/Group | Arm A (R2CHOP) | Arm B (RCHOP)
Number analyzed (Participants) | 145 | 135
proportion of participants | 0.97 [0.94 to 0.99] | 0.92 [0.87 to 0.95]

3. Secondary Outcome: Proportion of Patients With Complete Response
Description: Complete response is defined as complete disappearance of all detectable clinical evidence of disease, and disease-related symptoms if present prior to therapy.
Time Frame: Assessed every 3 months for 2 years, every 6 months for year 3, and then annually for years 4-10
Population: Evaluable (eligible and treated) patients
Measure: Number (90% Confidence Interval); unit: proportion of participants
Arm/Group | Arm A (R2CHOP) | Arm B (RCHOP)
Number analyzed (Participants) | 145 | 135
proportion of participants | 0.73 [0.66 to 0.79] | 0.68 [0.61 to 0.75]

4. Secondary Outcome: Overall Survival Rate at 3 Years
Description: Overall survival is defined as time from randomization to death or date last known alive. Overall survival rate at 3 years was calculated using the method of Kaplan Meier.
Time Frame: Assessed every 3 months for 2 years, every 6 months for year 3, and then annually for years 4-10
Population: Evaluable (eligible and treated) patients
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Arm A (R2CHOP) | Arm B (RCHOP)
Number analyzed (Participants) | 145 | 135
proportion of participants | 0.826 [0.765 to 0.892] | 0.751 [0.681 to 0.829]

5. Other Pre Specified Outcome: Impact of DLBCL Molecular Subtype on Outcome.
Time Frame: Assessed at baseline, every 3 months for 2 years, every 6 months for year 3, and then annually for years 4-10
Reporting Status: Not Posted

6. Other Pre Specified Outcome: Interim PET Scan Results in Relation to Treatment Outcome
Description: * To evaluate the association between the binary score of baseline SUV and PFS.
  * To evaluate the association between the binary score of % change in standard uptake value (SUVs) from PET3 to baseline and PFS.
Time Frame: Assessed every 3 months for 2 years, every 6 months for year 3, and then annually for years 4-10
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Assessed every 3 weeks while on treatment and for 30 days after the end of treatment, up to 10 years.
Description: Only patients who started protocol therapy are included in the analysis of adverse events. All registered patients are included in the analysis of all-cause mortality.
Arm/Group | Arm A (R2CHOP) | Arm B (RCHOP)
All-Cause Mortality (participants affected / at risk) | 36/173 | 43/176
Serious Adverse Events (participants affected / at risk) | 128/166 | 117/171
Other Adverse Events (participants affected / at risk) | 164/166 | 164/171
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A (R2CHOP) (N=166) | Arm B (RCHOP) (N=171)
Tinnitus (Ear and labyrinth disorders) | 1 | 0
Anemia (Blood and lymphatic system disorders) | 49 | 35
Febrile neutropenia (Blood and lymphatic system disorders) | 42 | 21
Leukocytosis (Blood and lymphatic system disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 2 | 0
Heart failure (Cardiac disorders) | 1 | 0
Left ventricular systolic dysfunction (Cardiac disorders) | 2 | 3
Pericarditis (Cardiac disorders) | 0 | 1
Restrictive cardiomyopathy (Cardiac disorders) | 1 | 0
Sinus bradycardia (Cardiac disorders) | 1 | 0
Cardiac disorders - Other, specify (Cardiac disorders) | 1 | 0
Edema limbs (General disorders) | 0 | 1
Fatigue (General disorders) | 17 | 11
Fever (General disorders) | 1 | 1
Infusion related reaction (General disorders) | 2 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 3 | 0
Toxic epidermal necrolysis (Skin and subcutaneous tissue disorders) | 1 | 0
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Colitis (Gastrointestinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 1 | 0
Diarrhea (Gastrointestinal disorders) | 10 | 1
Enterocolitis (Gastrointestinal disorders) | 1 | 0
Gastric hemorrhage (Gastrointestinal disorders) | 1 | 0
Gastric perforation (Gastrointestinal disorders) | 0 | 1
Ileal obstruction (Gastrointestinal disorders) | 0 | 1
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 | 0
Mucositis oral (Gastrointestinal disorders) | 5 | 3
Nausea (Gastrointestinal disorders) | 2 | 2
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Small intestinal perforation (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 2 | 0
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 1 | 1
Abdominal infection (Infections and infestations) | 1 | 0
Anorectal infection (Infections and infestations) | 1 | 0
Enterocolitis infectious (Infections and infestations) | 1 | 0
Lung infection (Infections and infestations) | 11 | 8
Pleural infection (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 11 | 10
Skin infection (Infections and infestations) | 2 | 0
Soft tissue infection (Infections and infestations) | 1 | 0
Upper respiratory infection (Infections and infestations) | 3 | 1
Urinary tract infection (Infections and infestations) | 6 | 2
Vaginal infection (Infections and infestations) | 1 | 0
Wound infection (Infections and infestations) | 0 | 1
Infections and infestations - Other, specify (Infections and infestations) | 5 | 4
Fall (Injury, poisoning and procedural complications) | 0 | 1
Spinal fracture (Injury, poisoning and procedural complications) | 1 | 0
Alanine aminotransferase increased (Investigations) | 1 | 1
Alkaline phosphatase increased (Investigations) | 1 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0
Blood bilirubin increased (Investigations) | 1 | 0
Creatinine increased (Investigations) | 1 | 0
Ejection fraction decreased (Investigations) | 2 | 1
Lymphocyte count decreased (Investigations) | 51 | 48
Lymphocyte count increased (Investigations) | 1 | 0
Neutrophil count decreased (Investigations) | 99 | 93
Platelet count decreased (Investigations) | 57 | 21
White blood cell decreased (Investigations) | 73 | 57
Alkalosis (Metabolism and nutrition disorders) | 0 | 1
Anorexia (Metabolism and nutrition disorders) | 4 | 2
Dehydration (Metabolism and nutrition disorders) | 6 | 4
Hyperglycemia (Metabolism and nutrition disorders) | 3 | 3
Hypoalbuminemia (Metabolism and nutrition disorders) | 2 | 1
Hypocalcemia (Metabolism and nutrition disorders) | 3 | 2
Hypokalemia (Metabolism and nutrition disorders) | 10 | 3
Hyponatremia (Metabolism and nutrition disorders) | 8 | 7
Hypophosphatemia (Metabolism and nutrition disorders) | 8 | 2
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 8 | 3
Muscle weakness right-sided (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal and connective tissue disorder - Other, spe (Musculoskeletal and connective tissue disorders) | 1 | 0
Aphonia (Nervous system disorders) | 1 | 0
Dizziness (Nervous system disorders) | 2 | 0
Peripheral motor neuropathy (Nervous system disorders) | 2 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 1 | 2
Stroke (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 5 | 3
Trigeminal nerve disorder (Nervous system disorders) | 0 | 1
Leukemia secondary to oncology chemotherapy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Treatment related secondary malignancy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Neoplasms benign, malignant and unspecified (incl cysts and (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Conjunctivitis (Eye disorders) | 1 | 0
Confusion (Psychiatric disorders) | 1 | 0
Delirium (Psychiatric disorders) | 0 | 1
Insomnia (Psychiatric disorders) | 0 | 2
Psychiatric disorders - Other, specify (Psychiatric disorders) | 1 | 0
Adult respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Acute kidney injury (Renal and urinary disorders) | 1 | 0
Renal calculi (Renal and urinary disorders) | 1 | 0
Hypertension (Vascular disorders) | 3 | 4
Hypotension (Vascular disorders) | 3 | 4
Thromboembolic event (Vascular disorders) | 6 | 4
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A (R2CHOP) (N=166) | Arm B (RCHOP) (N=171)
Anemia (Blood and lymphatic system disorders) | 144 | 134
Chills (General disorders) | 17 | 11
Edema limbs (General disorders) | 39 | 22
Fatigue (General disorders) | 126 | 135
Fever (General disorders) | 24 | 19
Infusion related reaction (General disorders) | 11 | 6
Pain (General disorders) | 5 | 10
Alopecia (Skin and subcutaneous tissue disorders) | 66 | 69
Dry skin (Skin and subcutaneous tissue disorders) | 10 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 12 | 6
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 16 | 2
Abdominal pain (Gastrointestinal disorders) | 16 | 13
Constipation (Gastrointestinal disorders) | 82 | 73
Diarrhea (Gastrointestinal disorders) | 58 | 42
Dry mouth (Gastrointestinal disorders) | 14 | 5
Dyspepsia (Gastrointestinal disorders) | 8 | 15
Mucositis oral (Gastrointestinal disorders) | 33 | 35
Nausea (Gastrointestinal disorders) | 76 | 48
Vomiting (Gastrointestinal disorders) | 32 | 18
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 9 | 6
Alanine aminotransferase increased (Investigations) | 12 | 13
Alkaline phosphatase increased (Investigations) | 15 | 7
Aspartate aminotransferase increased (Investigations) | 13 | 12
Blood bilirubin increased (Investigations) | 17 | 5
Creatinine increased (Investigations) | 8 | 11
Lymphocyte count decreased (Investigations) | 52 | 56
Neutrophil count decreased (Investigations) | 59 | 40
Platelet count decreased (Investigations) | 74 | 65
Weight loss (Investigations) | 28 | 26
White blood cell decreased (Investigations) | 60 | 34
Anorexia (Metabolism and nutrition disorders) | 47 | 46
Dehydration (Metabolism and nutrition disorders) | 9 | 17
Hyperglycemia (Metabolism and nutrition disorders) | 21 | 17
Hypoalbuminemia (Metabolism and nutrition disorders) | 34 | 25
Hypocalcemia (Metabolism and nutrition disorders) | 19 | 12
Hypokalemia (Metabolism and nutrition disorders) | 28 | 19
Hypomagnesemia (Metabolism and nutrition disorders) | 12 | 4
Hyponatremia (Metabolism and nutrition disorders) | 21 | 18
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 25 | 20
Myalgia (Musculoskeletal and connective tissue disorders) | 13 | 9
Pain in extremity (Musculoskeletal and connective tissue disorders) | 9 | 10
Dizziness (Nervous system disorders) | 26 | 24
Dysgeusia (Nervous system disorders) | 32 | 25
Headache (Nervous system disorders) | 19 | 14
Peripheral motor neuropathy (Nervous system disorders) | 12 | 14
Peripheral sensory neuropathy (Nervous system disorders) | 73 | 64
Insomnia (Psychiatric disorders) | 19 | 21
Cough (Respiratory, thoracic and mediastinal disorders) | 16 | 16
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 34 | 34
Hypertension (Vascular disorders) | 9 | 9
Hypotension (Vascular disorders) | 14 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-03-25): https://cdn.clinicaltrials.gov/large-docs/92/NCT01856192/Prot_SAP_000.pdf